CLINICAL TRIAL: NCT04950751
Title: An Observer-blind, Randomized, Controlled, Phase 2 Study to Evaluate the Immunogenicity and Safety of Clover Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2020S) in Adults
Brief Title: Immunogenicity and Safety of Adjuvanted SCB-2020S Vaccines in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decided to withdrawn the study as development strategy has changed
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2020-001
Record Dates: First submitted 2021-06-17; First posted 2021-07-06 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SCB-2020S Standard Dose (Experimental): Day 1 and 22: standard dose SCB-2020S with CpG 1018/alum adjuvant
  Interventions: Biological: candidate vaccine, SCB-2020S
- SCB-2020S Low Antigen Dose (Experimental): Day 1 and 22: low dose SCB-2020S with CpG 1018/alum adjuvant
  Interventions: Biological: candidate vaccine, SCB-2020S
- SCB-2020S Low Adjuvant Dose (Experimental): Day 1 and 22: standard dose SCB-2020S with low dose CpG 1018/alum adjuvant
  Interventions: Biological: candidate vaccine, SCB-2020S
- SCB-2020S Mixed Series (Experimental): Day 1 (Dose 1) standard dose SCB-2020S with CpG 1018/alum adjuvant and Day 22 Dose 2) standard dose SCB-2020S with alum adjuvant
  Interventions: Biological: candidate vaccine, SCB-2020S
- SCB-2019 (Active Comparator): Day 1 and 22: standard dose SCB-2019 with CpG 1018/alum adjuvant
  Interventions: Biological: candidate vaccine, SCB-2020S

INTERVENTIONS:
Biological: candidate vaccine, SCB-2020S — a recombinant SARS-Co-2 trimeric S-protein (from B.1.351 variant) subunit vaccine for COVID-19

SUMMARY:
This is a phase 2, randomized, controlled, observer-blind study to evaluate the immunogenicity and safety of different formulations of the investigational adjuvanted recombinant SARS-CoV-2 trimeric S-protein (from B.1.351 variant) subunit vaccine (SCB-2020S), when administered as 2-dose vaccination series 21 days apart to adults ≥ 18 years of age.

DETAILED DESCRIPTION:
Clover has developed a second candidate vaccine, SCB-2020S, that contains S protein from the dominant B.1.351 variant. The purpose of clinical study CLO-SCB-2020-001 is to assess the immunogenicity and safety of different formulations of the SCB-2020S compared to the prototype SCB-2019 vaccine, and to select a formulation of SCB-2020S for further clinical development. The protocol plans to enroll 150 participants. There will be 5 study arms and participants will receive two intramuscular (i.m.) injections, one at Day 1 and one at Day 22.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female ≥18 years of age
* 2. Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests and other study procedures.
* 3.Individuals are willing and able to give an informed consent, prior to screening
* 4. Healthy participants or participants with pre-existing medical conditions* who are in a stable medical condition. (*A stable medical condition is defined as disease not requiring significant change or hospitalization for worsening disease during the 3 months before enrollment.)
* 5. Female participants of childbearing potential may be enrolled in the study, if the participant has practiced adequate contraception for 30 days prior to vaccination and has a negative pregnancy test on the day of vaccination and has agreed to continue adequate contraception for 3 months after the last vaccination
* 6. Male participants must agree to employ acceptable contraception from the day of the first dose of the study vaccine until 6 months after the last dose of the study vaccine and also refrain from donating sperm during this period.

Exclusion Criteria:

* 1. Individuals with body temperature >37.5°C (axillary), or any acute illness at baseline (Day 1) or within 3 days prior to randomization. Participants meeting this criterion may be rescheduled within the relevant window. Febrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* 2. Individuals with laboratory-confirmed SARS-CoV-2 infection [as defined by reverse transcriptase polymerase chain reaction (RT-PCR) assay or Rapid COVID Antigen Test or an equivalent at Visit 1] or with history of COVID-19.
* 3. Individuals seropositive at Baseline for SARS-CoV-2.
* 4.Individuals who have received an investigational or authorized COVID-19 vaccine prior to Day 1, or plan to receive COVID-19 vaccine during the study period.
* 5. Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease [e.g., malignancy, human immunodeficiency virus (HIV) infection] or immunosuppressive/cytotoxic therapy (e.g., systemic corticosteroids, medications used for cancer chemotherapy, organ transplantation or to treat autoimmune disorders) within 3 months prior to Day 1.
* 6. Individuals with any progressive unstable or uncontrolled clinical conditions.
* 7. Individuals who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or during the study period.
* 8. Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction [e.g., anaphylaxis to any component of the study vaccines (CpG 1018, aluminum), or SCB-2020S/SCB-2019 components ].
* 9. Individuals who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
* 10. Individuals who have received any other investigational product within 30 days prior to Day 1 or intend to participate in another clinical study at any time during the conduct of this study.
* 11. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 21 days after the second vaccination.
* 12. Individuals with known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular injection.
* 13. Individuals who have received treatment with Rituximab or any other anti-CD20 monoclonal antibodies within 9 months prior to Day 1 or planned during the study period.
* 14. Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period.
* 15. Individuals with positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at Screening.
* 16. Individuals with safety laboratory test results (hematology, chemistry, and coagulation) with a toxicity score of Grade ≥2 at Screening (see Laboratory Manual for laboratory-specific normal ranges and associated toxicity grades). The inclusion of subjects with non-clinically significant (NCS) Grade 1 laboratory abnormalities is allowed based on the Investigator's discretion.
* 17. The subject has a reported or documented history of alcohol abuse or drug addiction or nonmedicinal recreational drug use (excluding nonprescription health supplements and herbal remedies) within 1 year before the planned day of dose administration.
* 18. The subject has a positive test result for drugs of abuse at Screening.
* 19. Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibodies to B.1.351 variant | Days 36
Proportion of subjects achieving seroconversion of SARS-CoV-2 neutralising antibodies to B.1.351 variant | Day 36
  Seroconversion rate (percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
Geometric mean fold rise (GMFR) of SARS-Cov-2 neutralising antibodies to B.1.351 variant | Day 36/Day 1

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibodies to Wuhan strain | Day 36
Proportion of subjects achieving seroconversion of SARS-CoV-2 neutralising antibodies to Wuhan strain | Day 36
  Seroconversion rate (percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
Geometric mean fold rise (GMFR) of SARS-Cov-2 neutralising antibodies to Wuhan strain | Day 36/Day 1
Geometric mean titer (GMT) of antibody titers specific to SCB-2019 antigen | Day 36
Proportion of subjects achieving seroconversion of antibodies specific to SCB-2019 | Day 36
  Seroconversion rate (percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
Geometric mean fold rise (GMFR) of antibodies specific to SCB-2019 | Day 36/Day 1
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibodies to B.1.351 variant | Day 205
Proportion of subjects achieving seroconversion of SARS-CoV-2 neutralising antibodies to B.1.351 variant | Day 205
  Seroconversion rate (percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
Geometric mean fold rise (GMFR) of SARS-Cov-2 neutralising antibodies to B.1.351 variant | Day 205/Day 1
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibodies to Wuhan strain | Day 205
Proportion of subjects achieving seroconversion of SARS-CoV-2 neutralising antibodies to Wuhan strain | Day 205
  Seroconversion rate (percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
Geometric mean fold rise (GMFR) of SARS-Cov-2 neutralising antibodies to Wuhan strain | Day 205/Day 1
Geometric mean titer (GMT) of antibody titers specific to SCB-2019 antigen | Day 205
Proportion of subjects achieving seroconversion of antibodies specific to SCB-2019 | Day 205
  Seroconversion rate (percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
Geometric mean fold rise (GMFR) of antibodies specific to SCB-2019 | Day 205/Day 1
Reactogenicity of the vaccines as indicated by the occurrence of solicited local reactions and solicited systemic adverse events. | 7 days after each dose
  Percentage of participants with local injection site reactions (pain, redness, swelling) and systemic adverse events (fatigue, headache, myalgia, arthralgia, loss of appetite, nausea, chills, and fever)
Safety of the vaccines in terms of the occurrence of unsolicited adverse events | Up to 21 days after second dose (Day 43)
  Percentage of participants with any adverse event other that those listed above as solicited adverse events
Safety of the vaccines in terms of the occurrence of medically attended adverse events (MAAEs), serious adverse events (SAEs), adverse events leading to discontinuation from study, and adverse events of special interest (AESI). | through study completion, an average of 7 months
  Percentage of participants with any adverse events in this category
Proportion of subjects with abnormal markers of hematology, biochemistry and coagulation parameters | Day 29